CLINICAL TRIAL: NCT02444377
Title: Impact of Varying High-intensity Interval Protocols on Cardiometabolic Risk Factors in Overweight/Obese
Brief Title: High-intensity Interval Training in Overweight/Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-1026
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2015-05

CONDITIONS: Obesity, Metabolically Benign
MeSH Terms: conditions — Obesity, Metabolically Benign | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-intensity interval -2min (Experimental): 5 bouts of 2 min cycling at varying intensities of VO2peak (80-100%) with 1 min recovery.
  Interventions: Behavioral: Interval training
- High-intensity interval -1min (Experimental): 10 bouts of 1 min cycling at 90% of VO2peak with 1 min rest periods
  Interventions: Behavioral: Interval training
- Control (No Intervention): No exercise

INTERVENTIONS:
Behavioral: Interval training
  Arms: High-intensity interval -1min; High-intensity interval -2min

SUMMARY:
Purpose: The purpose of this study would be to evaluate the effects of interval training on cardiovascular health, lipid profile and body composition in overweight and obese men and women.

A secondary purpose will be to compare lab based measurements of body composition [4-compartment model (4C)) with portable equipment [bioelectrical impedance spectroscopy (BIS) and ultrasound (US)]

Participants: Seventy-six men and women (age 18-55 yrs; BMI 25-45 kg/m2) will be randomly assigned to a high-intensity short interval group (SIT), high-intensity long interval group (HIT) or a control group (CON). Procedures (methods): Participants will be assessed for peak oxygen utilization (VO2peak), blood lipids, glucose and insulin levels. Body composition will also be measured using a 4C model, as measured from dual energy x-ray absorptiometry (DEXA), air displacement plethysmography (BodPod), and BIS, in comparison to US values. Participants assigned to either training group will undergo 3 weeks of interval training, 3 days per week. SIT will complete 10 bouts of a series of 1 min cycling with 1 min rest periods at 90% of the power output obtained during VO2peak;in comparison HIT will complete 5 bouts of the same protocol: 2 min bouts with 1 min recovery at varying intensities of VO2peak (80-100% power output).

ELIGIBILITY:
Inclusion Criteria:

* written and dated informed consent to participate in the study.
* willing and able to comply with the protocol.
* good health as determined by a health and exercise status questionnaire
* normal electrocardiogram (ECG), and physical.
* body mass index of 25-45 kg/m 2.
* has been cleared for participation by a physician (either study or personal).

Exclusion Criteria:

* participating in another clinical trial or have received an investigational product within thirty days prior to enrollment.
* has lost ten or more pounds during the previous three months and maintained the weight loss.
* significant history or current presence of untreated high blood pressure (BP) [systolic BP> 140 mmHg and/or diastolic BP> 90 mmHg], thyroid disease, tachyarrhythmia, heart disease, kidney disease, or liver disease. Subject currently suffers from/or has a known history of (or is currently being treated for) clinical depression or an eating disorder(s).
* has any medical condition or uses any medication, nutritional product, dietary supplement or program, which in the opinion of the investigator, might interfere with the conduct of the study or place the subject at risk.
* are identified as moderate to high risk individuals by the American College of Sports Medicine will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness (VO2peak) | 3 weeks

SECONDARY OUTCOMES:
Body Composition | 3 weeks
Blood Lipids | 3 weeks